CLINICAL TRIAL: NCT06427369
Title: Noninvasive Diagnosis of Lung Cancer With Radiolabeled hJAA-F11
Brief Title: An Investigational Scan (124I-hJAA-F11 PET/CT) for Diagnosing Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: prioritization
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I -1774023
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Extensive-stage Small-cell Lung Cancer; Limited-stage Small-cell Lung Cancer; Lung Non-Small Cell Carcinoma; Stage IIIA Lung Cancer; Stage IV Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic (Experimental): Patients receive 124I-hJAA-F11 IV on day 0. Patients then undergo PET/CT on day 1 (20-28 hours post 124I-hJAA-F11), day 2 (48-96 hours post 124I-hJAA-F11), day 5-6 (120-144 hours post 124I-hJAA-F11), and day 7-8 (168-192 hours post 124I-hJAA-F11). Patients also undergo FDG PET/CT during screening and undergo blood sample collection throughout the trial.
  Interventions: Other: Radioconjugate; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan; Procedure: Biospecimen Collection

INTERVENTIONS:
Other: Radioconjugate — 1241-hJAA-F11 IV administration
Procedure: Positron Emission Tomography — PET/CT Imaging
  Other Names: PET; PET SCAN
Procedure: Computed Tomography — PET/CT Imaging
  Other Names: CAT; CAT Scan
Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan — FDG PET/CT Imaging
  Other Names: FDG PET/CT
Procedure: Biospecimen Collection — Blood sample collection imaging
  Other Names: Biological Sample Collection

SUMMARY:
This phase I trial studies the side effects of 124I-hJAA-F11, and evaluates how well it works in diagnosing lung cancer. 124I-hJAA-F11 uses a known radioactive substance used in imaging called iodine 124 (124I). hJAA-F11 is an experimental (investigational) antibody that is currently being evaluated as a potential treatment for lung cancer. In animal studies, hJAA-F11 has shown anti-tumor activity against tumors bearing the Thomsen-Friedenreich antigen that is found in over 90% of lung cancers. 124I-hJAA-F11 has the 124I radioactive dye attached to this investigational antibody, which may be a potential tool for imaging-based diagnosis of lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and diagnostic efficacy of 124I-hJAA-F11 in detecting lung cancer.

SECONDARY OBJECTIVES:

I. To assess the development of anti-drug antibodies following administration of 124I-hJAAF11.

II. To characterize concordance in lesions characterized by 124I-hJAA-F11-based positron emission tomography/computed tomography (PET/CT) compared to standard of care FDG (fluorodeoxyglucose)-PET.

III. To perform exploratory biomarker analyses based on conventional tissue and liquid-based platforms.

OUTLINE:

Patients receive 124I-hJAA-F11 intravenously (IV) on day 0. Patients then undergo PET/CT on day 1 (20-28 hours post 124I-hJAA-F11), day 2 (48-96 hours post 124I-hJAA-F11), day 5-6 (120-144 hours post 124I-hJAA-F11), and day 7-8 (168-192 hours post 124I-hJAA-F11). Patients also undergo FDG PET/CT during screening and undergo blood sample collection throughout the trial.

After completion of the study intervention, patients are followed up at day 8-14, weeks 4 and 8, and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically diagnosed small cell lung cancer (SCLC; either extensive stage or limited stage) or non-small cell lung cancer (NSCLC; at least clinical stage IIIA according to the American Joint Cancer Committee [AJCC] 8th edition)
* Patients undergoing FDG-PET scan as standard of care testing.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection (exceptions allowed include patients on chronic antiviral or anti-bacterial medications without acute flares in the preceding 2 weeks), symptomatic congestive heart failure, unstable angina pectoris, Child-Pugh class C, dialysis-dependence, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3+ I-hJAA-F11 related adverse events | Up to 6 months after final PET/CT
  Incidence of severe adverse events will be graded according to CTCAE ver 5
Evaluate Diagnostic efficacy of I-hJAA-F11 | Within 30 days of final I/hJAA-f11 PET/CT
  uptake values for tumor and normal organs will be measured and tumor to normal orgrans background ratios will be obtained.

SECONDARY OUTCOMES:
Development of anti-drug antibodies | Up to approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace Dy, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center